CLINICAL TRIAL: NCT03728452
Title: Trophic Nutrition in Patients Submitted to High Flow Oxygen Therapy and / or Non Invasive
Brief Title: Trophic Nutrition in Patients Submitted to High Flow Oxygen Therapy and / or Non Invasive Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Hospital Universitario de Gran Canaria Doctor Negrín (Unknown); Hospital Universitario Fundación Jiménez Díaz (Other); Hospital Barbastro (Unknown); Hospital del Rio Hortega (Other); Hospital Universitario Infanta Cristina (Other); Hospital Universitario Ramon y Cajal (Other); University Hospital of Girona Dr. Josep Trueta (Network); Hospital Universitario Infanta Leonor (Other); Hospital Regional Universitario Carlos Haya (Other); Hospital de Cruces (Other); Hospital Universitario 12 de Octubre (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Virgen de la Concha (Unknown); Hospital Universitario de Torrevieja (Unknown); Complejo Hospitalario Universitario de Santiago (Other); Hospital Universitario Puerto Real (Other); Hospital Miguel Servet (Other); Hospital Universitario Severo Ochoa (Unknown); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Antonio Luis Blesa Malpica, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: 18/209-E
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Noninvasive Ventilation; Trophic Nutrition
Keywords: Trophic nutrition; high flow ventilation; noninvasive ventilation; mortality; complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Trophic Nutrition — According to previously published studies of Trophic Nutritions in critically ill patients, an energy goal of 20-30% estimated caloric needs of 20-30 kcal / kg and a protein intake of 1.2 to 2.0 g / kg / day of proteins will be established. at most 72 hours after the start of nutritional therapy.
  The rhythm of initiation and increase of enteral contributions will be at the discretion of each participating ICU. Prokinetic or parenteral nutrition (PN) complementary will not be used routinely, leaving its indication at the discretion of the responsible physician.
  A hyperproteic nutritional formula (10 g / 100 ml) will be used, with a caloric intake of 1.2 kcal / ml and a non-protein kcal / nitrogen ratio of 52: 1. TN will be administered over 23 hours each day by continuous infusion pump. The head of the patient's bed will rise above 30° as much as possible to reduce the risk of aspiration. The Gastric Residue Volume (GRV) will be measured every 24 hours.

SUMMARY:
The decision about the initiation of enteral nutrition therapy in critically ill patients with oxygen therapy needs with HFC and / or NIMV is a matter of debate at present. Despite the benefits associated with this practice in critically ill patients, the scarcity of clinical studies in patients with sufficient methodological quality, as well as the absence of specific recommendations on enteral nutrition therapy in this type of patient, generates controversy in the professionals involved in critical patient care.

DETAILED DESCRIPTION:
Ventilation and oxygenation of patients, even more in Intensive Care Units (ICUs), are in continuous development. The characteristics of patients, pathologies and diagnostic methods are constantly evolving. Among the main methods of ventilation and oxygenation that the investigators have are Non-invasive mechanical ventilation (NIMV) with face mask and high-flow cannula (HFC).

NIMV has represented an alternative in patients with failure to extubate, as an option before proposing a new reintubation. The ventilation with high flow has supposed an advance in the oxygenation of patients in situation of respiratory insufficiency, avoiding the intubation, and also has been a resource that allows the disconnection of the mechanical ventilator, reducing with it the time of mechanical support of the ventilation, There is a great amount of bibliography and a broad consensus on this aspect. Among the side effects widely studied, include bronchoaspiration, gastric insufflation, aerophagia and sialorrhea, which are usually well controlled with medical treatment.

The high flow ventilation consists of increasing the gas mixture, by releasing high oxygen and air flows, approximately up to 60 l/min, in modifiable proportions, so that positive pressures are achieved in the airway, facilitating the entry of this gas in the lung under spontaneous ventilation, with better oxygenation figures than conventional oxygen therapy methods. This positive pressure increase could be a facilitator of digestive intolerance either by air swallowing and gastric distension, or by promoting incontinence of the esophageal sphincters and thereby facilitating regurgitation and bronchoaspiration of the gastric contents.

NIMV consists of a ventilatory support applied without placement of endotracheal or pharyngeal devices, achieving increased alveolar ventilation by applying positive pressures throughout the airway through an interface (acting on the pressure gradient of the airway, to maintain an adequate gas exchange, impossible to achieve with spontaneous physiological ventilation). This positive pressure increase, as in ventilation with HFC, could also be an element that promotes digestive intolerance.

Patients in respiratory failure have a high level of metabolic stress that leads to a hypercatabolic situation and can not feed themselves for days, thus increasing the risk of malnutrition or worsening pre-existing malnutrition. This situation, as well as the development of negative energy balances in the critically ill patient, is associated with several complications, thus increasing morbidity and mortality, hospital stay and costs. The nutritional risk that this situation determines is high, which is why artificial nutrition therapy is justified. This nutritional therapy in spontaneous ventilation is usually attempted to be supplemented by oral feeding, but in patients who require artificial supports to aid in ventilation and oxygenation, it is not so easy to receive and tolerate adequate levels of caloric and protein intake. Enteral nutrition through the gastric route is frequently the method chosen for artificial nutritional therapy in patients with nutritional risk. This is due the advantages that the maintenance of the digestive tract in functional state will determine in the health of the patient, since the lack of nutrients in the lumen of the intestine can trigger a loss of the anatomical and functional integrity of the intestinal epithelium, with a rupture of the intestinal barrier that can favor, through a pro-inflammatory immune response, the evolution towards the multiple organ dysfunction syndrome.

ELIGIBILITY:
* INCLUSION CRITERIA:

  * Age ≥ 18 years.
  * Authorization to participate in the study through informed consent.
  * Patient with need of oxygen therapy with HFC and / or NIMV
  * NIMV or oxygen therapy time with HFC of at least 24 hours.
  * Expected survival over 72 hours.
  * Stay in ICU greater than or equal to 72 hours.
* EXCLUSION CRITERIA:

  * Age <18 years.
  * Denial of authorization to participate in the study.
  * Patient who does not require oxygen therapy with HFC and / or NIMV
  * Absolute contraindication for the onset of TN (active digestive hemorrhage, intestinal obstruction, etc.) or patients with non-functioning gastrointestinal tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in 3 spanish Intensive Medicine Units (ICU) in need of oxygen therapy with high-flow cannula and / or non-invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 2 year
  Numbers of patients death at 90 days

SECONDARY OUTCOMES:
Adverse effects | through study completion, an average of 2 year
  Numbers of Regurgitation, Vomits, Distension of Bronchoaspiration
Infections | through study completion, an average of 2 year
  numbers of all infections

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion para Investigación Biomedica Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Gay PC. Complications of noninvasive ventilation in acute care. Respir Care. 2009 Feb;54(2):246-57; discussion 257-8. PMID 19173756
- [Background] Liesching T, Kwok H, Hill NS. Acute applications of noninvasive positive pressure ventilation. Chest. 2003 Aug;124(2):699-713. doi: 10.1378/chest.124.2.699. PMID 12907562
- [Background] Thille AW, Contou D, Fragnoli C, Cordoba-Izquierdo A, Boissier F, Brun-Buisson C. Non-invasive ventilation for acute hypoxemic respiratory failure: intubation rate and risk factors. Crit Care. 2013 Nov 11;17(6):R269. doi: 10.1186/cc13103. PMID 24215648
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Background] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Background] Dvir D, Cohen J, Singer P. Computerized energy balance and complications in critically ill patients: an observational study. Clin Nutr. 2006 Feb;25(1):37-44. doi: 10.1016/j.clnu.2005.10.010. PMID 16321459
- [Background] Villet S, Chiolero RL, Bollmann MD, Revelly JP, Cayeux R N MC, Delarue J, Berger MM. Negative impact of hypocaloric feeding and energy balance on clinical outcome in ICU patients. Clin Nutr. 2005 Aug;24(4):502-9. doi: 10.1016/j.clnu.2005.03.006. PMID 15899538
- [Background] Deitch EA. Role of the gut lymphatic system in multiple organ failure. Curr Opin Crit Care. 2001 Apr;7(2):92-8. doi: 10.1097/00075198-200104000-00007. PMID 11373517
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Background] Mesejo A, Sanchez Alvarez C, Arboleda Sanchez JA; Spanish Society of Intensive Care Medicine and Coronary Units-Spanish Society of Parenteral and Enteral Nutrition (SEMICYUC-SENPE). [Guidelines for specialized nutritional and metabolic support in the critically ill-patient. Update. Consensus of the Spanish Society of Intensive Care Medicine and Coronary Units-Spanish Society of Parenteral and Enteral Nutrition (SEMICYUC-SENPE): obese patient]. Med Intensiva. 2011 Nov;35 Suppl 1:57-62. doi: 10.1016/S0210-5691(11)70012-2. Spanish. PMID 22309755
- [Background] Montejo JC, Minambres E, Bordeje L, Mesejo A, Acosta J, Heras A, Ferre M, Fernandez-Ortega F, Vaquerizo CI, Manzanedo R. Gastric residual volume during enteral nutrition in ICU patients: the REGANE study. Intensive Care Med. 2010 Aug;36(8):1386-93. doi: 10.1007/s00134-010-1856-y. Epub 2010 Mar 16. PMID 20232036
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Balogh Z, Offner PJ, Moore EE, Biffl WL. NISS predicts postinjury multiple organ failure better than the ISS. J Trauma. 2000 Apr;48(4):624-7; discussion 627-8. doi: 10.1097/00005373-200004000-00007. PMID 10780593
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Arabi YM, Aldawood AS, Haddad SH, Al-Dorzi HM, Tamim HM, Jones G, Mehta S, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Afesh L; PermiT Trial Group. Permissive Underfeeding or Standard Enteral Feeding in Critically Ill Adults. N Engl J Med. 2015 Jun 18;372(25):2398-408. doi: 10.1056/NEJMoa1502826. Epub 2015 May 20. Erratum In: N Engl J Med. 2015 Sep 24;373(13):1281. doi: 10.1056/NEJMx150028. PMID 25992505
- See also: Study ENVIN-HELICS. UCI infections — http://hws.vhebron.net/envin-helics/Help/Manual_2018.pdf